CLINICAL TRIAL: NCT05172440
Title: A Prospective Clinical Study on the Safety and Effectiveness of Tislelizumab Combined With Axitinib for Neoadjuvant Treatment of Clear Cell Renal Cell Carcinoma
Brief Title: A Study on the Safety and Effectiveness of Tislelizumab Combined With Axitinib for Neoadjuvant Treatment of ccRCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hongqian Guo (Other)
Responsible Party: Sponsor-Investigator, Hongqian Guo, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-RC-101
Record Dates: First submitted 2021-11-04; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-09

CONDITIONS: Neoadjuvant Therapy
Keywords: ccRCC; Neoadjuvant therapy; tislelizumab; axitinib
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- therapy group (Experimental): Subjects received axitinib 5 mg bid, 12 weeks, and tislelizumab 200 mg on the first day of the first week, 4th week, 7th week, and 10th week, and intravenous infusion. With 21 days as a treatment cycle, 4 cycles of treatment, namely 12 weeks. Axitinib was discontinued for 12 weeks after the completion of treatment, and surgery was performed 7 days later.
  Interventions: Drug: tislelizumab combined with axitinib

INTERVENTIONS:
Drug: tislelizumab combined with axitinib — Subjects received axitinib 5 mg bid, 12 weeks, and tislelizumab 200 mg on the first day of the first week, 4th week, 7th week, and 10th week, and intravenous infusion. With 21 days as a treatment cycle, 4 cycles of treatment, namely 12 weeks. Axitinib was discontinued for 12 weeks after the completion of treatment, and surgery was performed 7 days later.

SUMMARY:
This trial is a single-center clinical trial to evaluate the tumor shrinkage and safety of tislelizumab combined with axitinib in Neoadjuvant therapy of T2-T3N0M0 renal clear cell carcinoma

DETAILED DESCRIPTION:
The goal of the study is to use axitinib combined with tislelizumab in the Neoadjuvant therapy of T2-T3 N0M0 renal clear cell carcinoma to shrink tumors or tumor thrombi, reduce the complexity of surgery, and achieve kidney Partial resection or enucleation of renal tumors instead of kidney Partial resection, or unresectable renal tumors can be changed to resectable and improve the patient's prognosis.

The primary endpoint is the tumor shrinkage effect of tislelizumab combined with axitinib in Neoadjuvant therapy of T2-T3N0M0 renal clear cell carcinoma.

The secondary end point is

* The safety and downgrading rate of tislelizumab combined with axitinib in Neoadjuvant therapy of T2-T3N0M0 renal clear cell carcinoma；
* Two-year disease-free survival (DFS) of tislelizumab combined with axitinib in Neoadjuvant therapy of T2-T3N0M0 renal clear cell carcinoma；
* Explore biomarkers in tumor tissue and blood that may be related to the efficacy of neoadjuvant therapy and the prognosis of subjects;

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old
2. Imaging is consistent with T2-T3N0M0 renal cell carcinoma
3. Needle pathological biopsy is consistent with renal clear cell carcinoma
4. The subject intends to undergo radical nephrectomy or partial nephrectomy or renal tumor enucleation
5. ECOG 0-1 points
6. Normal hematopoiesis and organ function

   Hematopoietic function (no blood transfusion or blood products, no use of hematopoietic stimulating factors or other drugs to correct blood cells within 2 weeks before the first trial medication):

   Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet ≥100×109/L; Hemoglobin ≥9.0g/dL or ≥5.6mmol/L.

   Kidney function:

   Serum creatinine ≤ 1.5 times ULN, or serum creatinine> 1.5×ULN, the creatinine clearance rate is 60 mL/min; liver function: Total bilirubin≤1.5×ULN or total bilirubin>1.5×ULN but direct bilirubin is normal; AST and ALT≤2.5×ULN;

   Coagulation:

   International normalized ratio (INR) or prothrombin time (PT)≤1.5×ULN, and the activated part Thromboplastin time (aPTT)≤1.5×ULN; Left ventricular ejection fraction (LVEF) ≥50%
7. Able to sign informed consent
8. During the entire study period and within 3 months after the last administration, the subjects and their spouses are willing to use efficient contraceptive measures and not to donate sperm;
9. Understand and conduct visits, treatments, laboratory tests, and other research procedures as planned.

Exclusion criteria:

1. Previously received anti-tumor immunotherapy, including but not limited to cytokines (IL-2, IFN-α, etc.) and antibody drugs (anti-PD-1, PD-L1 or CTLA-4 antibodies, etc.);
2. Have previously received drug treatments targeting VEGF, VEGFR or mTOR, including but not limited to sunitinib, axitinib, sorafenib, pezopanib, cabotinib, lenvatinib, Bevacizumab or Iverolimus, etc.;
3. Participated in or currently participating in an experimental drug trial within 4 weeks before the first trial drug administration, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study; major surgery within 4 weeks before the first trial drug administration (Judgment by the investigator) or in the recovery period of surgery.
4. Receive Chinese medicine or Chinese patent medicine preparations with anti-tumor indications within 2 weeks before the administration of the first trial. Adrenal cortex hormones (>10 mg prednisone or equivalent drugs per day) or other immunosuppressive system treatments are required within 2 weeks before the first trial administration; those with >10 mg prednisone or equivalent drugs per day Inhalers, but those without active autoimmune diseases can participate in this study;
5. The toxicity has not been relieved after previous anti-tumor treatment, that is, it has not subsided to baseline, NCI-CTCAE 5.0 level 0~1 (except for hair loss), or the level specified in the inclusion/exclusion criteria. Irreversible toxicity (such as hearing loss) that is reasonably expected to not be aggravated by the study drug can participate in this study;
6. There are other malignant tumors that have progressed or need to be treated in the 5 years before enrollment (excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of breast, cervix or prostate);
7. There is a history of central nervous system (CNS) metastasis or the baseline imaging (MRI or CT) examination within 30 days before the first trial administration shows CNS metastasis;
8. Hypertension with poor control (systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥100mmHg) with a single drug;
9. The following cardiovascular events occurred in the 6 months before enrollment:

   1. Myocardial infarction
   2. Unstable angina
   3. Cardiovascular angioplasty or stent implantation
   4. Coronary artery/peripheral artery bypass grafting
   5. Grade III or IV congestive heart failure specified by the New York Heart Association
   6. Cerebrovascular accident or transient ischemic attack
10. QT interval (QTc) ≥480 msec corrected by heart rate (Bazett's formula);
11. A history of active bleeding or other severe bleeding within 30 days before enrollment, and a history of hemoptysis within 6 weeks before randomization;
12. Deep vein thrombosis or pulmonary embolism occurred within 6 months before enrollment;
13. Clinically significant gastrointestinal (GI) abnormalities, including:

    1. Malabsorption, total gastrectomy or any situation that may affect the absorption of oral drugs;
    2. Active ulcers that have been treated within the past 6 months;
    3. Active gastrointestinal bleeding (such as hematemesis, hematochezia or melena) within the past 3 months, and there is no evidence of recovery from endoscopic or colonoscopy;
    4. Suspected bleeding gastrointestinal metastatic lesions, inflammatory bowel disease, ulcerative colitis, gastrointestinal perforation or other gastrointestinal diseases that increase the risk of perforation;
14. A history of organ transplantation may require long-term adrenal cortex hormone therapy. Thyroid, adrenal or pituitary hypofunction that can be controlled only by hormone replacement therapy, type I diabetes, psoriasis or vitiligo that does not require systemic treatment, etc., can participate in this study;
15. Past or current (non-infectious) pneumonia/interstitial lung disease that requires adrenal cortex hormone therapy;
16. There are active infections that require systemic treatment, human immunodeficiency virus (HIV) infection (known HIV antibody positive), active HBV or HCV infection (HBsAg positive, or HBcAb positive but HBsAg negative). Additional DNA quantification tests can participate in this study if the result does not exceed the upper limit of the normal value of the research center laboratory; previous HCV infections have negative HCV RNA test results during the screening period, can participate in this study);
17. Live vaccines, including but not limited to mumps, rubella, measles, chickenpox/shingles (chickenpox), yellow fever, rabies, Bacille Calmette-Guerin (BCG) and typhoid vaccines within 30 days before enrollment, excluding inactivated viruses vaccine;
18. There is a history of severe drug allergy, including but not limited to antibody drugs and small molecule targeted drugs;
19. Known history of mental illness or drug abuse;
20. There is an unhealed wound;
21. Take it within 7 days before enrollment or expect to take it after enrollment, which is known as a strong CYP3A4/5 inhibitor and CYP3A4/5 inducer (including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, Rifampicin and Hypericum perforatum, etc.) or drugs that may cause arrhythmia (including but not limited to terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol and bep) Lee, etc.);
22. According to the judgment of the investigator, the subject has any medical history or current evidence of any disease, treatment or laboratory abnormality that may confuse the test results, interfere with the subject's participation in the entire trial, or do not meet the subject's best interest in participating in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-11-20 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate of tislelizumab combined with axitinib in neoadjuvant treatment of T2-T3N0M0 renal clear cell carcinoma | 7 days before surgery
  Objective response rate of tislelizumab combined with axitinib in neoadjuvant treatment of T2-T3N0M0 renal clear cell carcinoma

SECONDARY OUTCOMES:
The safety of tislelizumab combined with axitinib in neoadjuvant treatment of T2-T3N0M0 renal clear cell carcinoma | Follow-up period
  The safety of tislelizumab combined with axitinib in neoadjuvant treatment of T2-T3N0M0 renal clear cell carcinoma
Two-year disease-free survival (DFS) of tislelizumab combined with axitinib in neoadjuvant treatment of T2-T3N0M0 renal clear cell carcinoma | Three months to 2 years after surgery
  Two-year disease-free survival (DFS) of tislelizumab combined with axitinib in neoadjuvant treatment of T2-T3N0M0 renal clear cell carcinoma
Explore biomarkers in tumor tissue and blood that may be related to the efficacy of neoadjuvant therapy and the prognosis of subjects | Three months to 2 years after surgery
  The test content covers all exon regions of genes related to the prognosis, medication and development of kidney cancer, including homologous recombination repair (HRR) defect signaling pathways, WNT signal pathway , cell cycle pathway , MAPK signal pathway and chromosome remodeling signaling pathways
The downgrading rate of tislelizumab combined with axitinib in neoadjuvant treatment of T2-T3N0M0 renal clear cell carcinoma | Three months to 2 years after surgery
  The downgrading rate of tislelizumab combined with axitinib in neoadjuvant treatment of T2-T3N0M0 renal clear cell carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: shun zhang, Dr., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Hongqian Guo, Nanning, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No